CLINICAL TRIAL: NCT04573543
Title: The Role of Immune Semaphorins in NAFLD
Acronym: SepsisFAT
Status: Completed | Type: Observational
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: UHID-05
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2020-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Immune Response; Biomarkers; Liver Fibrosis; Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Non-alcoholic fatty liver disease: 120 patients diagnosed with NAFLD
  Interventions: Diagnostic Test: Evaluation of the degree of fibrosis and steatosis; Diagnostic Test: Screening for the components of metabolic syndrome; Diagnostic Test: Measurement of serum semaphorin concentrations; Diagnostic Test: Identification of semaphorin gene polymorphisms
- Controls: 40 healthy controls
  Interventions: Diagnostic Test: Evaluation of the degree of fibrosis and steatosis; Diagnostic Test: Screening for the components of metabolic syndrome; Diagnostic Test: Measurement of serum semaphorin concentrations; Diagnostic Test: Identification of semaphorin gene polymorphisms

INTERVENTIONS:
Diagnostic Test: Evaluation of the degree of fibrosis and steatosis — The degree of steatosis will be estimated using the controlled attenuation parameter (CAP), a method for grading steatosis by measuring the degree of ultrasound attenuation by hepatic fat using a process based on simultaneous transient elastography (TE) which measures the degree of fibrosis.
Diagnostic Test: Screening for the components of metabolic syndrome — Anthropometric measures including body mass index (BMI), waist circumference (WC), waist hip ratio (WHR), and waist height ratio (WHtR) will be measured in all patients.
  Results of the routine laboratory tests as part of the standard diagnostic procedure will be collected: bilirubin, AST, ALT, GGT, ALP, albumins, WBC, neutrophil-to-lymphocyte ratio, hemoglobin, platelet count, fasting glucose, triglycerides, cholesterol, HDL and LDL. Non-invasive scores of steatosis/fibrosis will be calculated (APRI, FIB4, NAFLD score). Patients will be screened for the components of metabolic syndrome.
Diagnostic Test: Measurement of serum semaphorin concentrations — Semaphorin concentration will be measured in patient sera by ELISA.
Diagnostic Test: Identification of semaphorin gene polymorphisms — Semaphorin genes will be sequenced to identify semaphorin gene polymorphisms associated with NAFLD.

SUMMARY:
To goal is to identify semaphorins that are associated with NAFLD and to investigate their relationship with variable degrees of steatosis and fibrosis.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common chronic liver disease associated with systemic changes in immune response. Semaphorins were recently recognized as one of the key regulators of immune responses; while some suppress immune cells activation, proliferation, and production of inflammatory cytokines, others stimulate immune responses. We have previously shown that semaphorins are associated with pathogenesis of viral hepatitis and progression of fibrosis. However, their role in NAFLD is unknown. The hypothesis of this project is that semaphorins are regulators of inflammation in patients with NAFLD. This study is designed as a prospective, non-interventional study. The main aims are: (1) to analyze serum concentration of semaphorins in patients with NAFLD; (2) to analyze tissue expression of semaphorins in patients with NAFLD; (3) to analyze semaphorin gene polymorphisms associated with NAFLD. Semaphorins could be a novel diagnostic and prognostic biomarker as well as targets for immune modulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with NAFLD according to current guidelines (AASLD, EASL)

Exclusion Criteria:

* Immunosuppression
* Malignancies
* Autoimmune diseases
* Pregnancy
* HIV
* Chronic viral hepatitis
* Presence of other chronic liver disease (hemochromatosis, Wilson's disease, toxic hepatitis, deficiency of alpha-1-antitrypsin, liver autoimmune disease)
* Consumption of alcohol > 20 g/day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 patients diagnosed with NAFLD and 40 healthy controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Detection of semaphorins in patients with NAFLD | 12 months
  Measurement of semaphorins concentration in serum of patients with NAFLD by enzyme-linked immunosorbent assay (ELISA)
Identification of semaphorin gene polymorphism in patients with NAFLD | 12 months
  Sequencing of semaphorin genes in patients with NAFLD using Sanger sequencing

SECONDARY OUTCOMES:
Staging of liver steatosis | 12 months
  The degree of steatosis will be estimated using the controlled attenuation parameter (CAP) in patients with NAFLD
Staging of liver fibrosis | 12 months
  The stage of liver fibrosis will be assessed by transient elastography (TE) in patients with NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Neven Papic, MD, PhD, Principal Investigator — University Hospital for Infectious Diseases Zagreb
Locations (1):
- University Hospital for Infectious Diseases Zagreb, Zagreb, Croatia

REFERENCES:
- [Result] Samadan L, Papic N, Mijic M, Knezevic Stromar I, Gasparov S, Vince A. Do Semaphorins Play a Role in Development of Fibrosis in Patients with Nonalcoholic Fatty Liver Disease? Biomedicines. 2022 Nov 23;10(12):3014. doi: 10.3390/biomedicines10123014. PMID 36551769